CLINICAL TRIAL: NCT02808000
Title: Evaluation of Suprapubic Noble Metal Alloy BIP Foley Catheter in the Prevention of Catheter-associated Urinary Tract Infections in Spinal Cord Injured Patients
Brief Title: BIP Foley in Prevention of CAUTI at Rehab Station
Acronym: CDOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bactiguard AB (Industry)
Collaborators: Rehab Station Stockholm (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 3686-2031-CDOC
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Complications; Catheter, Urinary Infection or Inflammation
MeSH Terms: conditions — Urinary Tract Infections; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (also called Group A ) (Active Comparator): Group 1/A will use standard catheter during the first ~6 months (observational period 1). Then the patients in this group will switch to the noble metal alloy urinary catheter (BIP Foley catheter of latex or silicone produced by Bactiguard AB) and be observed for another ~6 months (the second observational period).
  Interventions: Device: BIP Foley (latex) or BIP Foley -silicone; Device: Standard catheter
- Group 2 (also called Group B) (Experimental): Group 2/B will use the BIP Foley (latex or silicone) during the first ~6 months (observational period 1). Then the patients in this group will switch to the standard catheter and be observed for another ~6 months (the second observational period).
  Interventions: Device: BIP Foley (latex) or BIP Foley -silicone; Device: Standard catheter

INTERVENTIONS:
Device: BIP Foley (latex) or BIP Foley -silicone
  Other Names: Noble metal coated urinary catheters
Device: Standard catheter
  Other Names: Standard urinary catheter

SUMMARY:
This is a prospective, cross-over, randomized, controlled, partly blinded study evaluating safety and performance of noble metal alloy urinary Catheters (BIP Foley, Bactiguard AB) of both latex and silicone. The included patients are permanently catheterized spinal cord injured patients at the Spinalis clinic at Rehab station in Stockholm, Sweden.

Primary Outcome Measures:

• The primary objective is to evaluate the efficacy of long term suprapubic use of BIP Foley catheters, compared to the use of standard catheters for the same time period, on re-current symptomatic catheter associated urinary tract infection (CAUTIs).

Secondary Outcome Measures:

• to evaluate safety/performance of the catheter, i.e. antibiotic use, bacteriuria, bacteremia, urosepsis and ICU stay.

Exploratory Outcome Measures:

• assessment of levels of immunological markers in urine, urinary bacterial type and resistance pattern, catheter comfort, stability of the coating, and bacterial biofilm on the catheter surface after use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Patients with permanent suprapubic urethral catheter (Foley catheter) of latex or silicone
* At least 3 documented CAUTI infections during last year
* Spinal Cord Injured, changing catheters at Rehab Station every 10 weeks (+/- 2 weeks)

Exclusion Criteria:

* Children (˂18 years)
* Participating in other clinical trial(s) with exposure/treatment that could affect the outcome of the present study
* Stones (calculi) in the urinary tract (these patients can be included after the stones have been removed)
* Patients on antibiotic treatment (these patients can be included after the treatment is completed (+10 days of expectance))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Incidence of CAUTI | ~4 year observational time, the study has an open end and may be prolonged
  The frequency of CAUTI will be recorded and compared between the use of standard urinary catheter and BIP Foley (with noble metal coating)

SECONDARY OUTCOMES:
Incidence and typ of advese events | ~4 year observational time, the study has an open end and may be prolonged
  To assess and compare the frequency and type of adverse events and catheter related adverse events in the two arms
To compare ease of use of catheter by the nurse. Satisfaction assessed by ticking "easy" or "not easy" after each catheter exchange. | ~4 year observational time, the study has an open end and may be prolonged
  The coated and uncoated catheters will be compared with regards to number of easy catheterization.
Antibiotics type | ~4 year observational time, the study has an open end and may be prolonged
  To assess and compare any differences of type of antibiotics used for CAUTI in the two arms.
Antibiotics dose | ~4 year observational time, the study has an open end and may be prolonged
  To assess and compare any differences of antibiotic dose used for CAUTI in the two arms.
Antibiotics, number of treatment days | ~4 year observational time, the study has an open end and may be prolonged
  To assess and compare any differences of number of treatment days of antibiotics used for CAUTI in the two arms.
Incidence of spontaneous urinary and blood cultures and CRP blood | ~4 year observational time, the study has an open end and may be prolonged
  To asess and compare the spontaneous urinary and blood cultures and CRP blood in the two arms
Incidence of bacteruria, bacteremia, urosepsis and asymptomatic bacteremia | ~4 year observational time, the study has an open end and may be prolonged
  To asess and compare the incidence of bacteruria, bacteremia, urosepsis and asymptomatic bacteremiain the two arms

OTHER OUTCOMES:
To assess the stability of the coating during long term use, by measurement of the (i.e. Ag, Au and Pd) concentration in urine and in blood and on used catheters, | ~4 year observational time, the study has an open end and may be prolonged
  Urine and blood samples as well as used BIP Foley catheters, will be collected during the study visit, and the samples will be analysed with regards to metal concentrations (Ag, Au, and Pd).
To assess the comfort of BIP Foley Catheters. Comfort is measured by a questionnaire filled in by the patients. | ~4 year observational time, the study has an open end and may be prolonged
  The outcome of the questionnaire will be compared between the groups (standard versus coated catheter). The questions assess urine smell, appearance of the urine (i.e. colour), discomfort caused by the catheter, catheter blockage, discomfort at insertion/removal, and will be rated in a three-scale (not at all, little, much).
To asess inflammatory markers in urine of the patients and compare their levels between the groups. | ~4 year observational time, the study has an open end and may be prolonged
  Urine samples will be collected during the study visit, and will be analysed with regards to inflammatory markers. Inflammatory levels (e.g. cytokines IL-8 and microparticles) will be determined, and compared between the groups.
To assess bacterial type | ~4 year observational time, the study has an open end and may be prolonged
  The occurancy of bacterial strains in the two groups will be compared in urine samples collected at each study visit.
To assess bacterial resistance pattern. | ~4 year observational time, the study has an open end and may be prolonged
  The resistance pattern of present urinary bacteria in the two groups will be compared in urine samples collected at each study visit.
To assess and compare biofilm amount on the catheter surface. | ~4 year observational time, the study has an open end and may be prolonged
  Biofilm amount on the catheter surface of uncoated and coated catheters will be assessed and compared by using SEM. Amounts will be given as % biofilm covering the surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Åke Seiger, MD, Prof, Principal Investigator — Rehab Station Stockholm and Karolinska Institutet, Stockholm Sweden
Locations (1):
- Rehab Station Stockholm, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No